CLINICAL TRIAL: NCT02045030
Title: A Phase II Exploratory Study to Identify Biomarkers Predictive of Clinical Response to Aflibercept in Patients With Metastatic Colorectal Cancer Who Have Failed First-Line Therapy
Brief Title: Study to Identify Biomarkers of Clinical Response to Aflibercept in Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug (Aflibercept) no longuer available for the study
Sponsor: CR-CSSS Champlain-Charles-Le Moyne (Other)
Collaborators: Sanofi (Industry); Regeneron Pharmaceuticals (Industry); Quebec Clinical Research Organization in Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q-CROC-04
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic; colorectal; cancer; aflibercept; FOLFIRI
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — aflibercept; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept and FOLFIRI (Experimental): aflibercept and FOLFIRI
  Interventions: Drug: aflibercept + FOLFIRI

INTERVENTIONS:
Drug: aflibercept + FOLFIRI — Aflibercept (Sanofi and Regeneron) targets the Vascular endothelial growth factor (VEGF) pathway that is a composite decoy receptor based on VEGFR-1 and VEGFR-2 fused to an Fc segment of IgG1. In pre-clinical assessments, aflibercept results in stronger angiogenesis inhibition than bevacizumab, exhibiting at least 100-1000 times higher affinity to the circulating VEGFs. It is postulated that in vivo, the binding of these ligands to aflibercept results in the blockade of tumor angiogenesis along with pruning of existing tumor vascular elements and reduction of VEGF-driven vascular permeability. The expected outcome is reduced growth of primary and metastatic tumors by impeding the density of tumor vasculature and diminishing the abnormal leakiness of tumor vessels that supply matrix components to the cancer.
  Other Names: aflibercept; FOLFIRI

SUMMARY:
This is a Phase II multi-center exploratory study to identify biomarkers predictive of clinical response to aflibercept in patients with metastatic colorectal cancer who have failed first-line therapy, consisting of an oxaliplatin-containing regimen in combination with bevacizumab. Patients will consent to a needle core biopsy of a liver metastatic lesion prior to starting treatment and blood samples will be collected from study patients during treatment.

An exploratory pharmacoeconomic analysis will be performed to evaluate productivity loss, quality of life and resource utilization while on treatment with aflibercept.

DETAILED DESCRIPTION:
This is a Phase II multi-center exploratory study to identify biomarkers predictive of clinical response to aflibercept in patients with metastatic colorectal cancer who have failed first-line therapy, consisting of an oxaliplatin-containing regimen in combination with bevacizumab. Patients will consent to a needle core biopsy of a liver metastatic lesion prior to starting treatment. This study will be open primarily at sites conducting the Q-CROC-01 study (NCT00984048), in which colorectal cancer patients receiving standard first-line treatment undergo a biopsy of a liver metastatic lesion before treatment and at resistance. The post-first-line treatment biopsy will be used as the pre-treatment biopsy for this trial. For patients not participating in the Q-CROC-01 study, patients will be required to undergo a liver needle core biopsy of a metastatic lesion before study treatment.

Biopsies and blood samples will be collected from all study patients. An exploratory pharmacoeconomic analysis will be performed to evaluate productivity loss, quality of life and resource utilization while on treatment with aflibercept.

A total of 52 patients will be enrolled, primarily at centers participating in the Q-CROC-01 study. The trial will close enrolment when 42 evaluable pre-treatment tumor biopsy samples have been obtained. Accrual of the total patient population is estimated to take 24-36 months with the estimated start date being February 2014.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven adenocarcinoma of the colon or rectum, with at least one liver metastasis site available for biopsy.
2. Patients must have received only one prior chemotherapeutic regimen for metastatic disease. This prior chemotherapy must be an oxaliplatin containing regimen (in combination with bevacizumab). Patients who did not receive bevacizumab in their first-line treatment regimen may also be considered.
3. Metastatic disease that is not amenable to potentially curative treatment.
4. Measurable metastatic disease and evaluable disease.
5. ECOG 0 or 1.
6. Normal coagulation profile (PT, PTT, INR).
7. Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained.
8. Age ≥ 18 years.

Exclusion Criteria:

1. More than 1 prior chemotherapy regimen for metastatic colorectal cancer. Previous adjuvant FOLFOX based chemotherapy is allowed.
2. Relapse from adjuvant treatment within 6 month of completion of adjuvant chemotherapy.
3. Less than 42 days elapsed from prior major surgery to the time of registration.
4. Inadequate or unusable tissue as the only tissue available for biopsy.
5. Any of the following within 3 months of registration: Grade 3-4 gastrointestinal bleeding/hemorrhage, diverticulitis, pulmonary embolism, inflammatory or infections bowel disease, treatment resistant peptic ulcer disease, colitis, erosive esophagitis or gastritis, uncontrolled thromboembolic event.
6. Prior intolerance to bevacizumab due to toxicity.
7. Known dihydropyrimidine dehydrogenase (DPD) deficiency.
8. Gilbert's Syndrome.
9. Occurrence of deep vein thrombosis within 4 weeks, prior to registration.
10. Any of the following within 6 months prior to registration; myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack.
11. Contraindication to any of the components of the FOLFIRI chemotherapy regimen, as per investigators' judgement.
12. Inadequate bone marrow function as follows:

    * Absolute neutrophil count (ANC) < 1.5x 109/L
    * Platelet count < 100 x 109/L
    * Hemoglobin < 90 g/L
13. Inadequate liver function test:

    * Total bilirubin > 1.5 x ULN
    * Transaminases > 3 x ULN (if liver metastasis are present, 5 x ULN)
    * Alkaline phosphatase > 3 x ULN (if liver metastases are present, 5 x ULN)
14. Contraindication to aflibercept. Including:

    * Urine protein-creatinine ratio (UPCR) > 1 on morning spot urinalysis or proteinuria >500 mg/24-h
    * Serum creatinine > 1.5 x upper limit of normal (ULN). If creatinine 1.0 - 1.5 x ULN, creatinine clearance, calculated according to Cockroft-Gault formula, < 60 ml/min will exclude the patient.
    * History of uncontrolled hypertension, defined as blood pressure > 150/100 mgHG (grade ≥ 2 according to NCIC CTCAE v. 4.0), or systolic blood pressure > 180 mmHG when diastolic blood pressure < 90 mmHG, on at least 2 repeated determinations on separate days within 3 months prior to study enrollment.
    * Patients on anticoagulant therapy with unstable dose of warfarin and/or having an out-or-therapeutic range INR (>3) within the 4 weeks prior to study entry.
    * Evidence of clinically significant bleeding diathesis or underlying coagulopathy (eg. INR>1.5 without vitamin K antagonist therapy), non-healing wound.
15. Known active brain metastases or meningeal disease.
16. Female patients who are pregnant or breastfeeding.
17. Patients of reproductive potential (male and female) who do not agree to use an accepted form of contraception during the study period and up to 6 months following completion of study treatment.
18. Concurrent treatment with other anti-cancer therapy (palliative radiation is allowed but patients must have a metastatic site available for biopsy that has not been irradiated).
19. Known infection with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
A biomarker (in blood or tissue) that may be predictive of level of response to aflibercept | 3 years
  A biopsy from a liver metastasis will be taken at baseline for discovery of biomarkers that correlate with response to aflibercept. Genomic material (DNA and RNA) will be isolated from all biopsies. Batched analysis will be performed at the end of the study with the evaluable samples for multiplex biomarker discovery. Patient's biomarker status at baseline will be correlated with treatment effect on PFS and response (including response rate and disease control rate) to explore which biological targets may be particularly important in defining the appropriate treatment population for aflibercept.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Time from registration to progressive disease (up to 3 years)
  The time from the date of registration until the date of radiological disease progression assessed by RECIST 1.1 or until death due to any cause, even in the absence of radiological progression.
Response rate | 3 years
  Defined as complete response (CR) and partial response (PR)
Disease control rate | 3 years
  Defined as complete response (CR) + partial response (PR) + stable disease (SD).
Number of participants with adverse events | 3 years
  Assessment of safety profile of aflibercept in combination with FOLFIRI: report of Adverse Events according to the NCI's Common Toxicity Criteria version 4.0
The quality of life impact of treating with FOLFIRI in combination with Aflibercept | From date of registration until progression of disease assessed up to 36 months
  Quality of life will be evaluated by questionnaires completed by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Samson, MD, Principal Investigator — CSSS Champlain-Charles-Le Moyne
Locations (4):
- Canada (4):
  - CSSS Champlain-Charles-Le Moyne, Greenfield Park, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec

REFERENCES:
- [Background] Wang TF, Lockhart AC. Aflibercept in the treatment of metastatic colorectal cancer. Clin Med Insights Oncol. 2012;6:19-30. doi: 10.4137/CMO.S7432. Epub 2012 Jan 4. PMID 22253552
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Van Cutsem E, Tabernero J, Lakomy R, Prenen H, Prausova J, Macarulla T, Ruff P, van Hazel GA, Moiseyenko V, Ferry D, McKendrick J, Polikoff J, Tellier A, Castan R, Allegra C. Addition of aflibercept to fluorouracil, leucovorin, and irinotecan improves survival in a phase III randomized trial in patients with metastatic colorectal cancer previously treated with an oxaliplatin-based regimen. J Clin Oncol. 2012 Oct 1;30(28):3499-506. doi: 10.1200/JCO.2012.42.8201. Epub 2012 Sep 4. PMID 22949147